CLINICAL TRIAL: NCT00872911
Title: Nutrition and Exercise to Improve Protein Metabolism and Prevent Sarcopenia in Aging
Brief Title: Nutrition and Exercise for Sarcopenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08-085; 5R01AG030070 (NIH)
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; nutrition; aging; metabolism; exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Amino Acids; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nutritional supplement (Experimental)
  Interventions: Dietary Supplement: Amino acids
- Placebo + Exercise (Experimental)
  Interventions: Drug: Exercise
- Nutritional Supplement + Exercise (Experimental)
  Interventions: Dietary Supplement: Amino acids; Drug: Exercise
- Placebo (No Intervention)

INTERVENTIONS:
Dietary Supplement: Amino acids — mixed pure crystalline amino acids for human use (Ajinomoto), 15 g/d
  Arms: Nutritional Supplement + Exercise; Nutritional supplement
Drug: Exercise — progressive exercise training
  Arms: Nutritional Supplement + Exercise; Placebo + Exercise

SUMMARY:
The investigators' general hypothesis is that nutritional factors, including protein/energy malnutrition and/or an impaired response of muscle to nutrition, and inactivity play significant roles in developing sarcopenia, the involuntary loss of muscle mass and function with age. Therefore, age-specific prolonged interventions including nutritional manipulations and/or exercise may help to reduce, stabilize, or even reverse sarcopenia.

DETAILED DESCRIPTION:
Our preliminary studies indicate that, in older adults, muscle protein anabolism is normally stimulated by amino acids alone, but impaired when nutritional stimuli contain carbohydrate due to a relative insulin resistance of muscle protein synthesis. We have also found that amino acids are the most efficient nutrients for the acute stimulation of muscle protein anabolism and our pilot data suggest that they can also increase muscle mass in healthy older adults.

Inactivity is another likely contributor to sarcopenia. Exercise increases not only muscle protein synthesis,mass and strength, but also energy expenditure. Hence, exercise may improve the response of muscle to nutritional interventions in older subjects via increased energy requirements and food consumption, thereby allowing for achievement of true supplementation.

We will test the following specific hypotheses in older, community indwelling, sedentary subjects:

Using a factorial design we will address in older, community-indwelling, sedentary subjects the following hypotheses:

1. Nutritional supplementation with amino acids will improve muscle mass, strength, function, quality, and protein synthesis.
2. Progressive exercise training for 24 weeks will improve muscle mass strength,function, quality, perfusion, and protein metabolism.
3. Combined treatment with nutritional supplementation and progressive exercise training for 24 weeks will improve muscle mass, strength, function, quality, perfusion, and protein metabolism more than either intervention alone.

Our goal is to establish if specific interventions that can acutely increase muscle protein synthesis can also effectively translate into increased muscle mass and/or performance in older sedentary people, thus preventing frailty and promoting physical independence. To this end we will use stable isotope methodologies to measure muscle protein metabolism and contrast enhanced ultrasound to measure muscle perfusion, in order to determine if the treatments' acute effects can predict their chronic impact on muscle mass and function. We will also determine if chronic treatment leads to metabolic and/or vascular adaptations that may explain the measured changes in muscle mass and function.

ELIGIBILITY:
Inclusion Criteria:

1. age 65-85 yrs
2. ability to sign consent form (score >25 on the 30 item Mini Mental State Examination, MMSE)
3. stable body weight for at least 1 year (verified via medical records).

Exclusion Criteria:

1. physical dependence or frailty (impairment in any of the Activities of Daily Living (ADL), history of falls (≥2/year) or significant weight loss in the past year)
2. exercise training (≥2 weekly sessions of moderate-to-high intensity aerobic or resistance exercise)
3. significant heart, liver, kidney, blood or respiratory disease
4. peripheral vascular disease
5. diabetes or other untreated endocrine disease
6. active cancer
7. recent (within 6 months) treatment with anabolic steroids, or corticosteroids
8. alcohol or drug abuse
9. tobacco use (smoking or chewing, verified via medical records)
10. depression (>5 on the 15-item Geriatric Depression Scale (GDS))
11. malnutrition (BMI <20 kg/m2; hypoalbuminemia or hypotransferrenemia; protein intake<0.66 g/kg/day at run-in)
12. obesity (BMI>30 kg/m2).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-03; Primary Completion 2014-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Muscle mass | 6 months

SECONDARY OUTCOMES:
Muscle function | 6 months
muscle protein turnover | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elena Volpi, MD,PhD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- Sealy Center on Aging, University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Randolph AC, Markofski MM, Rasmussen BB, Volpi E. Effect of essential amino acid supplementation and aerobic exercise on insulin sensitivity in healthy older adults: A randomized clinical trial. Clin Nutr. 2020 May;39(5):1371-1378. doi: 10.1016/j.clnu.2019.06.017. Epub 2019 Jun 28. PMID 31307843
- [Derived] Markofski MM, Jennings K, Timmerman KL, Dickinson JM, Fry CS, Borack MS, Reidy PT, Deer RR, Randolph A, Rasmussen BB, Volpi E. Effect of Aerobic Exercise Training and Essential Amino Acid Supplementation for 24 Weeks on Physical Function, Body Composition, and Muscle Metabolism in Healthy, Independent Older Adults: A Randomized Clinical Trial. J Gerontol A Biol Sci Med Sci. 2019 Sep 15;74(10):1598-1604. doi: 10.1093/gerona/gly109. PMID 29750251